CLINICAL TRIAL: NCT06429007
Title: A Safety and Feasibility Trial Protocol of Metformin in Infants After Perinatal Brain Injury
Status: Enrolling by invitation | Phase: Phase 1 | Type: Interventional
Sponsor: Boston Children's Hospital (Other)
Responsible Party: Principal Investigator, Brian Kalish, Neonatologist, Assistant Professor of Pediatrics, Boston Children's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB-P00048370
Record Dates: First submitted 2024-05-07; First posted 2024-05-24 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Hypoxic-Ischemic Encephalopathy; HIE; Neurodevelopment; Infant Development
Keywords: HIE; metformin; Hypoxic-Ischemic Encephalopathy; Pharmacokinetic modeling; Neonates; Brain Injury
MeSH Terms: conditions — Hypoxia-Ischemia, Brain; Brain Injuries | interventions — Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Metformin Intervention (Experimental): Participants will complete a pre-study visit with baseline bloodwork including a complete blood count (CBC), liver and renal function, basic chemistry, glucose, and lactate. At this visit, parents will be taught how to administer metformin and given a 6-week supply (at 25% & 50% of the target dose for three weeks each) to minimize potential gastrointestinal upset. Parents will be educated on adverse effects and receive a diary to log dose administration and side effects. They will also be asked to perform at-home glucometer checks twice daily for 3 days post the dose escalation. After six weeks, participants will return for a study visit with repeat labs including assessing the levels of vitamin B12 and plasma metformin for measurement of pharmacokinetics. Parents will then receive a 6-week supply of metformin at the full dose (~25mg/kg) for 6 weeks. A final study visit will then occur following 12-weeks of metformin therapy, with repeat labs including plasma metformin levels.
  Interventions: Drug: Metformin

INTERVENTIONS:
Drug: Metformin — Metformin will be initiated at 25% of the target dose (4 mg/kg administered twice daily, total daily dose 8 mg/kg) for three weeks. In the absence of adverse effects, metformin dose will be escalated to 50% of the target dose (8 mg/kg administered twice daily for a total daily dose of 16mg/kg) for remaining 3 weeks to minimize potential gastrointestinal upset at higher doses. Parents will be documenting adverse events and performing glucometer checks twice a day for 3 days post dose escalation.
  Parents will then receive a 6-week supply of metformin at the target dose (16 mg/kg administered twice daily, total daily dose 32 mg/kg). Adverse events will be documented and glucometer checks will be performed twice a day for 3 days following dose escalation.

SUMMARY:
Infants with hypoxic-ischemic encephalopathy (HIE) are at high risk for neurodevelopmental impairment, despite current standards of care. Adjunctive treatments to promote brain repair are needed. The antidiabetic drug metformin has recently been recognized as a neurorestorative agent, but, to date, has not been used in infants. Herein, the investigator describes a clinical trial with the aim of demonstrating the safety and feasibility of metformin use to improve neurodevelopmental outcomes in infants with HIE.

ELIGIBILITY:
Inclusion Criteria:

* <6 months old at time of enrollment, and able to initiate study drug between 3 and 6 months old.
* Born > 35 weeks gestational age with a clinical diagnosis of HIE at birth, who receive therapeutic hypothermia.
* Post-hypothermia brain MRI with evidence of hypoxic-ischemic brain injury, based on the neuroradiology clinical report. Specifically, participants must have had evidence of a lactate peak by magnetic resonance spectroscopy and/or signal abnormalities by conventional (T1 and/or T2) or diffusion-weighted images consistent with hypoxic-ischemic pattern of injury.
* English- or Spanish-speaking families, as the parents/guardians will be responsible for documenting dose administrations and adverse events.

Exclusion Criteria:

* Known genetic or chromosomal disorder, and in the presence of congenital or acquired liver or kidney disease that might, in the opinion of the Principal Investigator (PI) or delegate, affect drug metabolism.
* Maternal use of metformin while actively breastfeeding.
* Infant weight below the 10th percentile based on WHO growth charts at the time of study drug initiation.
* Normal post-hypothermia brain MRI, without evidence of ischemic brain injury, based on the neuroradiology clinical report.
* Concomitant use of the following drugs: anti-diabetic drugs (insulin, sulfonylureas), steroids, diuretics (furosemide, chlorothiazide, spironolactone), diazoxide, beta blockers, ACE inhibitors, angiotensin II blockers, calcium channel blockers (including nifedipine), phenytoin, valproic acid, topiramate, cimetidine, corticosteroids, thyroid medications, sympathomimetics, carbonic anhydrase inhibitors, or any antibiotics.
* Any condition or diagnosis, that could in the opinion of the PI or delegate, interfere with the participant's ability to comply with study instructions, might confound the interpretation of the study results, or put the participant at risk.

Ages: 3 Months to 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Estimated)
Dates: Start 2025-10-01 (Actual); Primary Completion 2028-01-01 (Estimated); Study Completion 2029-03-01 (Estimated)

PRIMARY OUTCOMES:
Safety profile of kidney function | 12 weeks
  A renal function panel (chem 10 with renal function) will be performed prior to the initiation of therapy and at all subsequent study visits.
Safety profile of liver function | 12 weeks
  A liver function test (LFT) will be performed prior to the initiation of therapy and at all subsequent study visits.
Recruitment feasibility | 12 weeks
  To assess feasibility, the number of eligible patients will be compared to the number of patients who consent to participate in the study.

SECONDARY OUTCOMES:
Validity of neonatal model of metformin pharmacokinetics | 12 weeks
  Plasma metformin levels will be analyzed by investigators with whole blood obtained at study visits.

CONTACTS AND LOCATIONS:
Overall Officials: Brian Kalish, MD, Principal Investigator — Boston Children's Hospital
Locations (1):
- Boston Children's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hutchinson AM, Pais R, Endginton AN, Pilon B, MacDonald JM, MacDonald ME, Lewis T, Offringa M, Kalish BT. Safety and feasibility trial protocol of metformin in infants after perinatal brain injury. BMJ Paediatr Open. 2025 Aug 24;9(1):e002784. doi: 10.1136/bmjpo-2024-002784. PMID 40850908